CLINICAL TRIAL: NCT02333656
Title: Improved Management of Patients With Hip and Knee Osteoarthritis in Primary Health Care
Brief Title: Management of Hip and Knee Osteoarthritis in Primary Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Nina Osteras, Researcher, Diakonhjemmet Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 229079
Record Dates: First submitted 2015-01-04; First posted 2015-01-07 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Usual care. The participants enrolled in the control period will receive OA treatment as it is currently offered in primary health care services.
- Intervention group (Experimental): New OA model. Health professionals attend an interactive workshop, implementation of international recommendations for OA care, multidiciplinary collaboration
  Interventions: Other: New OA model

INTERVENTIONS:
Other: New OA model — The general practitioners and the physiotherapists will attend an inter-active workshop and deliver osteoarthritis care in line with international recommendations for osteoarthritis treatment. The general practitioner will refer eligible patients to treatment by physiotherapists at "Healthy Living Center" or by physiotherapists in private practice. This treatment will include a standardized patient education program followed by structured exercise program with individual adjustments. The general practitioner will schedule a follow-up after the 12-week treatment and will receive a treatment report from the physiotherapist.
  Arms: Intervention group

SUMMARY:
Previous research has shown that the osteoarthritis care for persons with hip or knee osteoarthritis in Norway has a potential for improvement as the provided care may not necessarily reflect evidence-based guideline recommendations. This study will determine if a new model for integrated osteoarthritis (OA) care in primary health care will result in improved quality of osteoarthritis care and health benefits for the patients (reduced pain and body weight, increased function and activity level) among patients with hip and/or knee osteoarthritis. Further, this study will examine if the new model reduce the number of unnecessary referrals to Magnetic Resonance Imaging (MRI) and to orthopaedic surgeons in secondary care, and if it increases the number of referrals to physiotherapy treatment and the number of discharge reports from the physiotherapists to the referring general practitioner.

DETAILED DESCRIPTION:
A new model for integrated care for patients with hip and/or knee osteoarthritis (OA) in primary care will be developed and implemented. The purpose of the model is to improve quality of OA care in primary health care services by increasing the collaboration between health care professionals and across health care levels, providing an integrated care and a patient pathway, and facilitating an active and healthy lifestyle among individuals with OA. This implementation study represents a collaborative study between six municipalities and a hospital department aiming to fulfill the intentions of the Norwegian Health Care Coordination Reform. The main aim of the present study is to implement and perform process and effect evaluations of this new model for integrated OA care. The study design will be a cluster randomized controlled trial with a stepped wedge design. Six neighboring municipalities will constitute the six clusters, which will switch from control (current OA care) to intervention phase (new OA model) in a randomized order. All municipalities start the trial simultaneously and act as controls until the point in time they are randomized to crossover from control to intervention, and all municipalities have implemented the intervention by the end of inclusion. The method consists of two parts; 1) Identification of barriers/facilitators + development of the model and interventions, 2) Implementation of the new model (interactive workshops) with process and effect evaluations. Participants will be general practitioners and physiotherapists in primary care as well as people with hip or knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Activity-related hip and/or knee pain/complaints AND
* Clinical signs and symptoms corresponding to hip and/or knee OA OR radiologically diagnosed OA OR Registered in the medical journal with the ICPC codes L89 (osteoarthritis of the hip), L90 (osteoarthritis of knee), L91 (osteoarthritis not classified elsewhere), L13 (hip symptoms/complaints), L15 (knee symptoms/complaints) and/or L20 (joint symptoms/complaints not classified elsewhere).

Exclusion Criteria:

* Total hip or knee replacement in the actual joint(s) and no pain/complaints in the other hip or knee joint(s)
* Inflammatory rheumatic diseases (e.g. rheumatoid arthritis, spondyloarthritis)
* Malignant illness or other major conditions (i.e unstable cardiovascular disorders or lung disease, dementia) that restrict the ability to adhere to the recommended OA treatment
* Do not understand the Norwegian language

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Osteoarthritis Quality Indicator questionnaire | 6 months
  Patient reported achievement of quality indicators for osteoarthritis care

SECONDARY OUTCOMES:
Pain | 6 months
  Pain level in hip/knee past week
Joint stiffness | 6 months
  Stiffness in the hip/knee past week
Global function | 6 months
  Hip/knee function in the past week
Patient global assessment of the OA disease | 6 months
Patient Acceptable Symptom State (PASS) | 6 months
Hip/knee function, quality of living subscale | 6 months
  Function (Knee injury and Osteoarthritis Outcome Score ADL subscale/ Hip disability and Osteoarthritis Outcome Score OoL subscale (K/HOOS)
Physical activity level | 6 months
  An index based on self-reported frequency, intensity, duration of physical activity
Daily sitting | 6 months
  Daily hours in sitting position
Satisfaction with the care provided | 6 months
Health related quality of life (EQ-5D) | 6 months
Self-reported body weight | 6 months
Health care use, medication use and sick leave | 6 months
Adverse events | Up to 1 year
Health professionals' knowledge, attitude and behavior in OA care | Pre- and post-workshop + 6 months post-workshop
Referrals to orthopaedic surgeons | Up to 1 year
  Number of referrals to secondary care that does not lead to scheduled joint surgery
Referrals to MRI | Up to 1 year
  Number of referrals to MRI for OA assessment
Number of referrals to physiotherapy treatment | Up to 1 year
Discharge reports from physiotherapists | Up to 1 year
  Number of discharge reports from PTs at FLSs/ private practice to the referring GP
Arthritis Self-efficacy Scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kåre Hagen, Prof., Study Director — Project administrator/Research director; Nina Østerås, PhD, Principal Investigator — Researcher
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

REFERENCES:
- [Derived] Osteras N, Aas E, Moseng T, van Bodegom-Vos L, Dziedzic K, Natvig B, Rotterud JH, Vlieland TV, Furnes O, Fenstad AM, Hagen KB. Longer-term quality of care, effectiveness, and cost-effectiveness of implementing a model of care for osteoarthritis: A cluster-randomized controlled trial. Osteoarthritis Cartilage. 2024 Jan;32(1):108-119. doi: 10.1016/j.joca.2023.10.003. Epub 2023 Oct 13. PMID 37839506
- [Derived] Moseng T, Dagfinrud H, van Bodegom-Vos L, Dziedzic K, Hagen KB, Natvig B, Rotterud JH, Vlieland TV, Osteras N. Low adherence to exercise may have influenced the proportion of OMERACT-OARSI responders in an integrated osteoarthritis care model: secondary analyses from a cluster-randomised stepped-wedge trial. BMC Musculoskelet Disord. 2020 Apr 13;21(1):236. doi: 10.1186/s12891-020-03235-z. PMID 32284049
- [Derived] Osteras N, Moseng T, van Bodegom-Vos L, Dziedzic K, Mdala I, Natvig B, Rotterud JH, Schjervheim UB, Vlieland TV, Andreassen O, Hansen JN, Hagen KB. Implementing a structured model for osteoarthritis care in primary healthcare: A stepped-wedge cluster-randomised trial. PLoS Med. 2019 Oct 15;16(10):e1002949. doi: 10.1371/journal.pmed.1002949. eCollection 2019 Oct. PMID 31613885
- [Derived] Moseng T, Dagfinrud H, Osteras N. Implementing international osteoarthritis guidelines in primary care: uptake and fidelity among health professionals and patients. Osteoarthritis Cartilage. 2019 Aug;27(8):1138-1147. doi: 10.1016/j.joca.2019.03.010. Epub 2019 May 8. PMID 31075423
- [Derived] Osteras N, van Bodegom-Vos L, Dziedzic K, Moseng T, Aas E, Andreassen O, Mdala I, Natvig B, Rotterud JH, Schjervheim UB, Vlieland TV, Hagen KB. Implementing international osteoarthritis treatment guidelines in primary health care: study protocol for the SAMBA stepped wedge cluster randomized controlled trial. Implement Sci. 2015 Dec 2;10:165. doi: 10.1186/s13012-015-0353-7. PMID 26631224